CLINICAL TRIAL: NCT06401161
Title: Study on the Effect of 3T Pu'er Tea in Regulating Glucose and Lipid Metabolism
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Longgang District People's Hospital of Shenzhen (Other)
Responsible Party: Principal Investigator, Chen Yuhua, Chief physician, Longgang District People's Hospital of Shenzhen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LonggangDPHS
Record Dates: First submitted 2022-11-22; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Overweight; Obesity
Keywords: Pu' er Tea; glucose and lipid metabolism; intestinalflora
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The recommended method for consuming 3T Pu-erh tea is as follows: according to individual preferences, once a day, 8 g/time, or twice a day, 4 g/time, using a 300 mL stew cup; Steep the tea in 200 mL of boiling water for 60-90 seconds and consume. The tea can be brewed multiple times, replacing regular water intake. Ensure that the entirety of the liquid in the cup is consumed during each session.
  Interventions: Other: 3T Pu'er tea
- Control group (Placebo Comparator): The recommended method for consuming traditional Pu-erh tea is as follows: according to individual preferences, once a day, 8 g/time, or twice a day, 4 g/time, using a 300 mL stew cup; Steep the tea in 200 mL of boiling water for 60-90 seconds and consume. The tea can be brewed multiple times, replacing regular water intake. Ensure that the entirety of the liquid in the cup is consumed during each session.
  Interventions: Other: 3T Pu'er tea

INTERVENTIONS:
Other: 3T Pu'er tea — Two types of Pu-erh tea with different levels of theabrownin content.
  Other Names: Traditional Pu'er tea

SUMMARY:
To study the effect of Pu'er tea in overweight / obese patients with blood glucose or abnormal lipid metabolism. Compared with the effect of two Pu'er tea with different tea fuscin content in improving glucose and lipid metabolism, to investigate the mechanisms of bile acid metabolism and intestinal flora regulation.

In a prospective randomized controlled clinical study, 90 patients were divided into study group (3T Pu'er tea group, 45 patients) and control group ( traditional Pu'er tea group,45 patients). Before and after the treatment(0day, 12 weeks, 52 weeks) patients' markers of glucose and lipid metabolism were examined and compared.

ELIGIBILITY:
Inclusion Criteria:

The A、B should be simultaneously met, or combined with the C、D、E.

1. 18-65 years, priority for patients over 30 years;
2. Overweight / obese patients: BMI ≥24 kg/m2.
3. Or combined with nonalcoholic fatty liver disease: determined by the hospital MRI nuclear magnetic quantification;
4. Or combined with dyslipidemia: blood total cholesterol TC≥6.4mmol/L or blood total triglyceride TG≥2.0mmol/L or blood low-density lipoprotein LDL-C≥3.1mmol/L;
5. Or with abnormal blood glucose:

   * Impaired fasting glucose, IFG: fasting blood glucose was 6.1~<7.0mmol/L,and 2 hours after 75g oral blood glucose tolerance test(OGTT) <7.8mmol / L.
   * Impaired glucose tolerance, IGT: the fasting blood glucose was <6.1mmol/L and 2 hours after 75gOGTT was 7.8~ <11.1 mmol / L;
   * IFG with IGT: patients with both IFG and IGT;
   * Patients with type 2 diabetes: random blood glucose 11.1mmol/L or fasting glucose of 7.0 mmol/L or 2 hours after OGTT.

Exclusion Criteria:

1. Type 2 diabetes and insulin injections or oral hypoglycemic drugs and other special types of diabetes.
2. For women during pregnancy or lactation or with allergies;
3. Patients treated with any hypoglycemic drugs and insulin injections; regular or planned patients taking drugs that may affect glucose and lipid metabolism (as judged by clinicians, such as diet pills, lipid-lowering drugs) and liver protection drugs (as judged by clinicians);
4. Patients with severe cardiovascular diseases, cerebrovascular diseases, liver, kidney, and hematopoietic diseases;
5. Combined with other infectious diseases, such as hepatitis A, hepatitis B, hepatitis C, and acquired immunodeficiency syndrome;
6. Take probiotics, prebiotics, antioxidants and fish oil nutrient supplements within 3 months;
7. Current smokers and regular drinking (excluding social drinkers only);
8. Yogurt intake within 1 week before the first visit and antibiotics within 3 months;
9. Drink strong tea regularly;
10. Participate in other clinical trials within 3 months;
11. Unable not cooperate with the investigator for other reasons.
12. Unfit for the researcherr.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood lipids | 0week
  Blood lipids were detected by the Roche COBAS C702 biochemical analyzer.
Blood lipids | 6weeks
  Blood lipids were detected by the Roche COBAS C702 biochemical analyzer.
Blood lipids | 12weeks
  Blood lipids were detected by the Roche COBAS C702 biochemical analyzer.
Blood lipids | 52weeks
  Blood lipids were detected by the Roche COBAS C702 biochemical analyzer.
Blood glucose | 0week
  Blood glucose were detected by the Roche COBAS C702 biochemical analyzer.Normal reference range：Fasting Blood Glucose 3.9-6.1 mmol/L.
Blood glucose | 6weeks
  Blood glucose were detected by the Roche COBAS C702 biochemical analyzer.Normal reference range：Fasting Blood Glucose 3.9-6.1 mmol/L.
Blood glucose | 12weeks
  Blood glucose were detected by the Roche COBAS C702 biochemical analyzer.Normal reference range：Fasting Blood Glucose 3.9-6.1 mmol/L.
Blood glucose | 52weeks
  Blood glucose were detected by the Roche COBAS C702 biochemical analyzer.Normal reference range：Fasting Blood Glucose 3.9-6.1 mmol/L.
Hepatic fat fraction indicators | 0week
  Siemens 3.0T medical MRI equipment was applied for MAFLD diagnosis and fat quantitative assessment.
Hepatic fat fraction indicators | 12weeks
  Siemens 3.0T medical MRI equipment was applied for MAFLD diagnosis and fat quantitative assessment.
Hepatic fat fraction indicators | 52weeks
  Siemens 3.0T medical MRI equipment was applied for MAFLD diagnosis and fat quantitative assessment.
Intestinal flora detection | 0week
  Polymerase Chain Reaction amplification was carried out in the v1-v9 variable region of the 16S rRN gene using universal primer (27F-1492R), and sequencing was conducted in the Illumina novaseq platform. The 16S rRNA amplicon sequence was processed using QIIME2. VSEARCH software was adopted to splice, filter, and remove chimeras from the original sequence to obtain the effective sequences. Clustering was performed according to the 99% similarity of the sequences to obtain the operational taxonomic units (OTU). Based on the Silva NR99 132 database, the representative sequences were analyzed and annotated. The OTU list was generated. The abundance and classification of all OTUs in the samples were recorded.
Intestinal flora detection | 12weeks
  Polymerase Chain Reaction amplification was carried out in the v1-v9 variable region of the 16S rRN gene using universal primer (27F-1492R), and sequencing was conducted in the Illumina novaseq platform. The 16S rRNA amplicon sequence was processed using QIIME2. VSEARCH software was adopted to splice, filter, and remove chimeras from the original sequence to obtain the effective sequences. Clustering was performed according to the 99% similarity of the sequences to obtain the operational taxonomic units (OTU). Based on the Silva NR99 132 database, the representative sequences were analyzed and annotated. The OTU list was generated. The abundance and classification of all OTUs in the samples were recorded.
Intestinal flora detection | 52weeks
  Polymerase Chain Reaction amplification was carried out in the v1-v9 variable region of the 16S rRN gene using universal primer (27F-1492R), and sequencing was conducted in the Illumina novaseq platform. The 16S rRNA amplicon sequence was processed using QIIME2. VSEARCH software was adopted to splice, filter, and remove chimeras from the original sequence to obtain the effective sequences. Clustering was performed according to the 99% similarity of the sequences to obtain the operational taxonomic units (OTU). Based on the Silva NR99 132 database, the representative sequences were analyzed and annotated. The OTU list was generated. The abundance and classification of all OTUs in the samples were recorded.

SECONDARY OUTCOMES:
Creatinine | 0week
  Creatinine was detected by the Roche COBAS C702 biochemical analyzer. Normal reference range：Creatinine: Female 44-97umol/L, Male 53-106umol/L.
Creatinine | 12weeks
  Creatinine was detected by the Roche COBAS C702 biochemical analyzer. Normal reference range：Creatinine: Female 44-97umol/L, Male 53-106umol/L.
Creatinine | 52weeks
  Creatinine was detected by the Roche COBAS C702 biochemical analyzer. Normal reference range：Creatinine: Female 44-97umol/L, Male 53-106umol/L.
Bone densitometry | 0 week
  The bone mineral density of the axial skeleton (L1-4 vertebrae, left femoral neck, total hip) of the subjects was measured in g/cm2 using a dual-energy X-ray absorptiometry (coefficient of variation <1%) from Hologic, USA.
Bone densitometry | 52 weeks
  The bone mineral density of the axial skeleton (L1-4 vertebrae, left femoral neck, total hip) of the subjects was measured in g/cm2 using a dual-energy X-ray absorptiometry (coefficient of variation <1%) from Hologic, USA.
Alanine aminotransferase | 0week
  Creatinine was detected by the Roche COBAS C702 biochemical analyzer. Normal reference range：Alanine aminotransferase: 0-40U/L.
Alanine aminotransferase | 12weeks
  Creatinine was detected by the Roche COBAS C702 biochemical analyzer. Normal reference range：Alanine aminotransferase: 0-40U/L.
Alanine aminotransferase | 52weeks
  Creatinine was detected by the Roche COBAS C702 biochemical analyzer. Normal reference range：Alanine aminotransferase: 0-40U/L.

CONTACTS AND LOCATIONS:
Locations (1):
- Longgang District People's Hospital of Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Study Protocol, Clinical Study Report are to be shared with other researchers.